CLINICAL TRIAL: NCT04276506
Title: Comparison of the Effect of Music and Giving Information on the Patient Care Who Undergoing Coronary Angiography
Brief Title: Effect of Information Given and Music on the Care of Patient Who Will Undergo Coronary Angiography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EasternMUU
Record Dates: First submitted 2020-01-27; First posted 2020-02-19 (Actual); Last update posted 2020-09-28 (Actual); Status verified 2020-01

CONDITIONS: Anxiety State; Invasive Procedure
Keywords: Anxiety; Coronary Angiography; Nursing; Music; Visual Information; Physiological parameters
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- information booklet group (Experimental): information session before the coronary angiography
  Interventions: Other: information group
- music group (Experimental): music session before the coronary angiography
  Interventions: Other: music group
- control group (No Intervention): No information or music session before the coronary angiography

INTERVENTIONS:
Other: music group — to reduce anxiety, some selected music pieces will have patients listened by headset.
  Arms: music group
Other: information group — A visual information booklet which is prepared by the researchers will be used
  Arms: information booklet group

SUMMARY:
Today, due to the increasing frequency of cardiovascular diseases the number of coronary angiography performed has also risen. This invasive procedure has an effect on patients which causes anxiety. Its important to determine of the level of anxiety so experienced nurses carried out various interventions to reduce anxiety.

This study aims to determine the effect of listening music and getting information on the level of anxiety and vital signs of the patients who are planned to undergo coronary angiography.

For this purpose, calming music which is suitable for the heart rhythm and booklets which is prepared with various visuals will be used. In the study, apart from a control group that routine clinical procedures will be applied, there will be two more groups which are called as music and information groups. Patients' participation in these groups will be distributed randomly by computer.

DETAILED DESCRIPTION:
The patients will be included to this study who will undergo coronary angiography first time and admitted to hospital by appointment.

Inserting IV canulla, taking and recording vital signs, and informing about angiography are routine procedures for patients who are admitted to hospital for coronary angiography. These procedures will also be applied to the patient groups involved in the study.

Patients will be assigned to the groups in accordance with the randomization table. After explaining the purpose and method of the study to the patients, their consent will be obtained.In this experimental study all datas will be collected by Descriptive Characteristics Form, Vital Findings Follow-Up Form and The State-Continuity Anxiety Inventory.

Vital Signs Follow-Up Form will be recorded according to patients' findings, such as heart rate per minute, blood pressure as mmHg and respiratory rate per minute both before and after angiography.

The State-Continuity Anxiety Inventory will be applied before angiography to determine the anxiety level of the patients. After the angiography, the state anxiety inventory will be repeated.The information group; A visual information booklet which is prepared by the researcher will be used. In the booklet; Information about coronary arteries, angiography laboratory features, patient preparation procedure and post-procedure are explained with various visuals. The booklet which contains researchers telephone numbers will be given to patients, when they come to hospital to get an angiography appointment. The patients will be asked to read the booklet until the day of angiography. If patients need to ask some questions, they will be able to reach the researchers within specified hours.

The Music group; A soothing type of music including five kinds sounds of nature which suitable for heart rate was selected and recorded on MP3. When they arrive hospital for angiography they will be explained how to use MP3 player and headset in the room. All music stored on the MP3 player will be played to the patient for five to ten seconds. They will be asked to choose their preferred music. The patient will listen the music which is chosen for 30 minutes via headset. In order to prevent contamination, disposable ear cups will be used for each patient.

ELIGIBILITY:
Inclusion Criteria:

* adult
* patients who undergoing coronary angiography first time
* able to speak and understand turkish
* people informed clearly by the investigator

Exclusion Criteria:

* having any hearing and visual problems
* being on psychiatric medications
* emergency cases
* patient under legally protection

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2019-11-10 (Actual); Primary Completion 2020-01-10 (Actual); Study Completion 2020-03-10 (Actual)

PRIMARY OUTCOMES:
State anxiety level | 1 day
  Use of the State-Trait Anxiety Inventory (STAI) to assess the level of anxiety

SECONDARY OUTCOMES:
heart rate | 1 day
  beats per minute
respiratory rate | 1 day
  breaths per minute
blood pressure | 1 day
  mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Handan Sezgin, Assist Prof., Study Director — Eastern Mediterranean University Health Science Faculty; Nurdan Yıldız, Msc, Principal Investigator — Eastern Mediterranean University Health Science Faculty
Locations (1):
- EMU Health Science Faculty, Famagusta, Cyprus

IPD SHARING:
Plan to Share IPD: No